CLINICAL TRIAL: NCT07055555
Title: Disrupted Connections: The Impact of Acute Stress on Memory Integration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nevada State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2501-0392; 5P20GM103440 (NIH)
Record Dates: First submitted 2025-06-05; First posted 2025-07-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Stress; Control Condition
Keywords: acute stress; memory; memory integration; cognitive maps
MeSH Terms: interventions — Psychological Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Stress Condition (Experimental): Participants randomized to the acute stress condition will complete the Trier Social Stress Test (TSST), a validated experimental method for inducing acute psychosocial stress. This condition will allow for us to evaluate our primary hypothesis.
  Interventions: Behavioral: Acute Stress
- Non-Stress Control Condition (Sham Comparator): Participants randomized to the non-stress control condition will complete a non-stressful task designed to parallel the structure of the Trier Social Stress Test without eliciting acute stress.
  Interventions: Behavioral: Non-Stress Control Task

INTERVENTIONS:
Behavioral: Acute Stress — Participants randomized to the acute stress condition will complete the Trier Social Stress Test (TSST), a validated experimental method for inducing acute psychosocial stress. The TSST consists of a brief anticipation period followed by a 5-minute mock job interview and a 5-minute surprise mental arithmetic task, performed in front of a neutral panel of judges in professional attire.
  Other Names: Trier Social Stress Test
  Arms: Acute Stress Condition
Behavioral: Non-Stress Control Task — Participants randomized to the control condition will complete a non-stressful task designed to parallel the structure of the Trier Social Stress Test without eliciting acute stress. They will have a brief anticipation period followed by a 5-minute description of their typical day or favorite hobby. This task is conducted without an evaluative panel, minimizing the potential for stress or anxiety.
  Arms: Non-Stress Control Condition

SUMMARY:
The goal of this study is to better understand how stress impacts people's ability to learn across their experiences and link new information to what they already know. The investigators will compare performance on a memory task between stressed and non-stressed participants. This memory task requires people to integrate knowledge across learning experiences (think: having to "connect the dots", draw inferences, and generalize your knowledge to new situations and scenarios). Cortisol, the brain's primary stress hormone, will be measured at multiple points throughout the study to measure stress levels. The investigators hypothesize that:

1. Stress will disrupt performance on the memory task by interfering with memory processes that enable linking of related memories.
2. Higher cortisol levels, which reflect a greater stress response, will relate to greater deficits in memory performance across participants.

This research has broad implications for understanding how stress impacts the ability to learn and retain new information, particularly in high-stress environments like schools and workplaces. Additionally, this work may provide insights into the cognitive difficulties experienced by individuals with psychiatric disorders, where stress can worsen memory and learning challenges.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* aged 18-35 years
* speak fluent English
* have normal or corrected-to-normal vision

Exclusion Criteria:

* individuals who are pregnant
* exercise within 1 hour of the study session
* smoking within 1 hour of the study session
* consuming drugs or alcohol within 1 hour of the study session

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Performance on A-C inference trials in the Paired Associative Inference Task | During the participant's study visit, anticipated 1-2 hours
  Performance on A-C inference trials of the memory task assesses memory integration across overlapping learning experiences.

SECONDARY OUTCOMES:
Performance on directly learned pairs (A-B and B-C) in the Paired Associative Inference Task | During the participant's study visit, anticipated 1-2 hours
  Performance on directly learned pairs (A-B and B-C) evaluates basic associative memory.

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Fernandez, PhD, Neuroscience, Principal Investigator — Nevada State University
Locations (1):
- Nevada State University, Henderson, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, including demographic and outcome measures, will be made available to qualified researchers upon request after publication of findings. Data will be shared under a data use agreement via a secure repository such as Open Science Framework (OSF).